CLINICAL TRIAL: NCT05670002
Title: Nutrition Intervention of Complementary Milk Feeding to Improve Linear Growth of at Risk and Stunted Children Aged Between 12-36 Months
Brief Title: Nutrition Intervention of Complementary Milk Feeding to Improve Linear Growth of at Risk and Stunted Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FrieslandCampina (Industry)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Moana
Record Dates: First submitted 2022-12-21; First posted 2023-01-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: At Risk or Stunted Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Other): Taking milk supplement
  Interventions: Dietary Supplement: Milk supplement

INTERVENTIONS:
Dietary Supplement: Milk supplement — Children will take the milk supplement for a period of 6 months. During the intervention, anthropometry data, Zinc Protoporphyrin levels, dietary intake, any illness will be recorded.

SUMMARY:
This is a non-randomized open label 6 months intervention study that aims to assess the effectiveness of consuming milk daily for 6 months will improve the linear growth rate of children aged 12-36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Malaysian child
2. Boys and girls between the age of 12 and 36 months
3. Length-for-age z score (LAZ) <-1.5 SD and > -3 SD according to the WHO Growth standard
4. Weight-for-age z score WAZ <1.0 SD and > -3 SD
5. Parents and/or legal guardian who can speak and read Malay or English language
6. Written informed consent from parents and/or legal guardian
7. Child who are apparently healthy with no obvious on-going infection and no history of chronic illness.
8. Child with no physical and/or mental illness
9. Parents and/or legal guardian who owns a mobile phone or smart phone
10. Mothers who have ever received breastfeeding counselling from a qualified breastfeeding counsellor.

Exclusion Criteria:

1. Child with zinc protoporphyrin (ZnPP) value of >65 (at either -T3 or T0)
2. Clinical symptoms of iron deficiency as examined by Doctor even with zinc protoporphyrin (ZnPP) value between 40-64
3. Child with severe acute malnutrition, other chronic diseases or any congenital disorder or deformity
4. Child with an ongoing episode of diarrhoea or a history of persistent diarrhoea in the past month
5. Child with history of cow's milk allergy/intolerance to milk
6. Child who is already taking multivitamins, including iron, before enrolled to the study
7. Child who is taking breastmilk as part of the diet

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Linear growth | 6 months
  Change in LAZ/HAZ z-score from baseline to after 6 months of intervention

SECONDARY OUTCOMES:
Growth velocity | 9 months
  Compare growth velocity between 3 months pre- to first 3 months and 6 months post intervention
Zinc Protoporphyrin (ZnPP) levels | 9 months
  Any change in ZnPP levels pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Jan Jan Mohamed, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- School of Health Sciences, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No